CLINICAL TRIAL: NCT01996956
Title: Prediction of Fluid Responsiveness by NICOM (Non-invasive Cardiac Output Monitoring) in Children With Congenital Heart Disease After Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Ph.D, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: H-1303-114-478
Record Dates: First submitted 2013-11-17; First posted 2013-11-27 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Fluid Responsiveness
Keywords: stroke volume variation,; cardiac output,; fluid responsiveness,; noninvasive cardiac output monitor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Volume loading (Other)
  Interventions: Other: volume expansion

INTERVENTIONS:
Other: volume expansion — fluid loading of 10 ml/kg colloid or blood product

SUMMARY:
The purpose of this study is to evaluate the ability of fluid responsiveness by stroke volume variation value of NICOM(Noninvasive cardiac output monitor)system during congenital cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* congenital cardiac surgery
* < 6 years old
* who were required the evaluation by transesophageal echocardiography

Exclusion Criteria:

* right heart failure
* supported by more than 2 inotropic agents
* reduced kidney function
* any valvar stenosis
* moderate or severe tricuspid regurgitation
* single ventricle

Ages: 1 Day to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2013-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
stroke volume index | before and after volume loading (20 min)
  Volume loading was performed for 20 minutes. Stroke volume measured before and after volume expansion using transesophageal echocardiography. And, stroke volume variation of NICOM monitor was recorded before fluid loading.

SECONDARY OUTCOMES:
Cardiac index | before and after fluid loading (20 min)
  Cardiac index measured by transesophageal echocardiography and NICOM monitor were compared before and after fluid loading for 20 min.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, MD, PhD, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul national university hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee JH, No HJ, Song IK, Kim HS, Kim CS, Kim JT. Prediction of fluid responsiveness using a non-invasive cardiac output monitor in children undergoing cardiac surgery. Br J Anaesth. 2015 Jul;115(1):38-44. doi: 10.1093/bja/aev109. Epub 2015 Apr 29. PMID 25926311